CLINICAL TRIAL: NCT07349147
Title: Thulium Fiber Laser Enucleation of the Prostate: Learning Curve and Functional Outcomes - A Prospective Study
Acronym: ThuFLEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muharrem Baturu (Other)
Responsible Party: Sponsor-Investigator, Muharrem Baturu, Assistant Professor, University of Gaziantep
Organization: University of Gaziantep (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2026/01
Record Dates: First submitted 2026-01-08; First posted 2026-01-16 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Prostate Hyperplasia; Thulium Fiber Laser; Laser Prostate Enucleation
Keywords: ThuFlep; Prostate enucleation; learning curve; laser enucleation
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Thulium Fiber Laser Enucleation of the Prostate (ThuFlEP) Group (Experimental): All patients in this study group will undergo Thulium Fiber Laser Enucleation of the Prostate (TfLEP) for the treatment of symptomatic Benign Prostatic Hyperplasia (BPH). The surgical procedure involves using a 60-watt Thulium Fiber Laser (TFL) system to enucleate the prostatic adenoma in a retrograde or antegrade fashion. Following enucleation, the adenoma is removed from the bladder using a mechanical morcellator. The study will monitor the surgeon's performance from the first consecutive case to evaluate the learning curve (measured by operative efficiency) and assess functional outcomes (IPSS, Qmax, and Quality of Life) at post-operative intervals of 1, 3, and 12 months.
  Interventions: Device: Thulium Fiber Laser (TFL) Enucleation

INTERVENTIONS:
Device: Thulium Fiber Laser (TFL) Enucleation — Surgical enucleation of the prostate using TFL technology to achieve complete removal of the transition zone adenoma, aiming for symptomatic relief and improvement in urinary flow.

SUMMARY:
The aim of this prospective study is to evaluate the learning curve and functional outcomes of Thulium Fiber Laser Enucleation of the Prostate (TfLEP) performed by a single surgeon. The study focuses on surgical efficiency, safety (complication rates), and the improvement of lower urinary tract symptoms (LUTS) and quality of life over a 12-month follow-up period.

DETAILED DESCRIPTION:
Thulium Fiber Laser (TFL) is an emerging technology in the field of laser prostatectomy. While Holmium Laser Enucleation (HoLEP) is well-established, the learning curve and long-term functional stability of TFL need further prospective validation. This study will involve the first [Insert Number, e.g., 100] consecutive cases of TfLEP. The "Learning Curve" will be analyzed using Cumulative Sum (CUSUM) analysis of enucleation efficiency and operative time. Functional outcomes will be assessed via IPSS, Qmax, and IIEF-5 scores at baseline and post-operative intervals (1, 3, and 12 months).

ELIGIBILITY:
Inclusion Criteria:

* Patients with symptomatic Benign Prostatic Hyperplasia (BPH) refractory to medical treatment.
* Prostate volume > [e.g., 40] ml.
* Patients providing written informed consent for the prospective follow-up

Exclusion Criteria:

* Neurogenic bladder dysfunction.
* Active urinary tract infection at the time of surgery.

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2025-10-01 (Actual); Study Completion 2026-01-01 (Actual)

PRIMARY OUTCOMES:
Learning Curve Competency | 12 month
  The point at which the surgeon achieves a stable enucleation efficiency (grams of tissue/minute) and a significant reduction in operative time.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Gaziantep,, Gaziantep, Gazi̇antep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes